CLINICAL TRIAL: NCT03764800
Title: The Prevalence of Micronutrient Deficiency in Early School-age Children and Its Correlation With Eating Behavior, Dietary Habits, Development, Physical Activity, Nutritional Status and Health Status
Brief Title: The Prevalence of Micronutrient Deficiency in Early School-age Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsun-Chin Chao, Attending Physician, Chang Gung Memorial Hospital
Other Study IDs: 201801719A3
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Micronutrient Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aim to assess the prevalence of deficiency in micronutrients in early school-age children and its correlation with picky eating behavior, physical activity, nutritional status, and health status.

DETAILED DESCRIPTION:
A structured questionnaire is used to conduct a cross-sectional descriptive study of 250 early school-age children aged 4-7 years (<7 years old) in Taiwan. Data collection would include: demographics, food preferences, eating behavior, body weight and height, body mass index (BMI), physical activity, records of medical illness, peripheral cell blood count, serum values of ferritin and micronutrients (iron, zinc, copper). Data from children define as picky or non-picky eaters base on parental' questionnaire responses, are analyzed and compared using standard statistical tests. The correlations among eating behavior, dietary habits, development, physical activity, nutritional status, and health status, and micronutrient deficiency are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 4-7 years old (<7 years old) school-age children, legal representatives willing to sign the consent form and fill in the questionnaire

Exclusion Criteria:

* At the time of the enrollment, there is an acute infection (respiratory, gastrointestinal or urinary tract), and there are organic diseases (heart, lung, brain, hepatobiliary, kidney, endocrine metabolic disease or heredity).

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This cross-sectional descriptive study uses a structured questionnaire to elicit information from parents in Taiwan who are early school-age children aged 4-7 years (<7 years old). Participants are recruited from clinic in Chang Gung Children's medical center, Chang Gung Memorial Hospital. A total of 250 participants who meet the eligibility criteria are enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-12-05 (Estimated)

PRIMARY OUTCOMES:
Change serum concentrations of Hb (g/dL) may be found in children's serum | On the day of enrollment
  Change serum concentrations of Hb (g/dL) may be found in children with picky eating behavior, low quality of development, inadequacy of physical activity, undernutrition, and poor health status.
Change serum concentrations of ferritin (ng/ mL) may be found in children's serum | On the day of enrollment
  Change serum concentrations of ferritin (ng/ mL) may be found in children with picky eating behavior, low quality of development, inadequacy of physical activity, undernutrition, and poor health status.
Change serum concentrations of iron (μg/dL), zinc (μg/dL), and copper (μg/dL) may be found in children's serum | On the day of enrollment
  Change serum concentrations of iron (μg/dL), zinc (μg/dL), and copper (μg/dL) may be found in children with picky eating behavior, low quality of development, inadequacy of physical activity, undernutrition, and poor health status.

CONTACTS AND LOCATIONS:
Overall Officials: Hsun-Chin Chao, A.P., Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No